CLINICAL TRIAL: NCT00280657
Title: Multicenter, Double-blind, Double-dummy, Randomized Parallel Group Study to Evaluate the Safety and Efficacy of SH D 00659 E for 6 Treatment Cycles in Female Patients With Acne Papulopustulosa in Comparison to SH D 00659 G and Placebo.
Brief Title: Study on Safety and Efficacy of an Oral Contraceptive in Treating Acne Papulopustulosa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 91299; 307760
Record Dates: First submitted 2006-01-20; First posted 2006-01-23 (Estimated); Last update posted 2023-06-06 (Actual); Status verified 2023-06

CONDITIONS: Acne Vulgaris
Keywords: Acne papulopustulosa
MeSH Terms: conditions — Acne Vulgaris | interventions — Cyproterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm 1 (Experimental)
  Interventions: Drug: Valette
- Arm 2 (Active Comparator)
  Interventions: Drug: Diane
- Arm 3 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Valette — 1 tablet 0.030 mg ethinylestradiol / 2 mg dienogest + 1 placebo tablet daily for 21 days followed by a 7-day tablet-free interval, oral administration for 6 cycles
  Arms: Arm 1
Drug: Diane — 1 tablet 0.035 mg ethinylestradiol / 2 mg cyproterone acetate + 1 placebo tablet daily for 21 days followed by a 7-day tablet-free interval, oral administration for 6 cycles
  Arms: Arm 2
Drug: Placebo — 2 placebo tablets daily for 21 days followed by a 7-day tablet-free interval, oral administration for 6 cycles
  Arms: Arm 3

SUMMARY:
The purpose of the study is to determine safety and efficacy of an oral contraceptive in treating acne papulopustulosa.

DETAILED DESCRIPTION:
The study has previously been posted by Schering AG, Germany. Schering AG, Germany has been renamed to Bayer Schering Pharma AG, Germany.Bayer Schering Pharma AG, Germany is the sponsor of the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with mild to moderate facial papulopustular acne

Exclusion Criteria:

* Contraindication against use of hormonal contraceptives

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1326 (Actual)
Dates: Start 2004-03-10 (Actual); Primary Completion 2005-05-21 (Actual); Study Completion 2005-05-21 (Actual)

PRIMARY OUTCOMES:
Change in lesions | 6 months

SECONDARY OUTCOMES:
ISGA | 6 months
Parameters of safety and tolerability | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (43):
- Czechia (9):
  - Chomutov
  - Čáslav
  - Kutná Hora
  - Louny
  - Olomouc
  - Prague
  - Slaný
  - Svitavy
  - Ústí nad Labem
- Poland (6):
  - Grudziądz
  - Lodz
  - Lublin
  - Poznan
  - Warsaw
  - Wroclaw
- Russia (5):
  - Korolyov
  - Moscow
  - Moskva
  - Petrozavodsk
  - Saint Petersburg
- Slovakia (5):
  - Banská Bystrica
  - Bratislava
  - Kosice-Saca
  - Košice
  - Nitra
- Ukraine (18):
  - Alchevs'k
  - Chernivtsi
  - Dnipropetrovsk
  - Donetsk
  - Ivano-Frankivsk
  - Kharkiv
  - Kiev
  - Kyiv
  - Luhansk
  - Lviv
  - Makiivka
  - Odesa
  - Poltava
  - Rivne
  - Simferopol
  - Ternopil
  - Uzhhorod
  - Zaporizhzhia